CLINICAL TRIAL: NCT06480357
Title: A Giant Myelolipoma, Management by Laparoscopy.
Brief Title: A Giant Myelolipoma.
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Huber Díaz Fuentes, Dr., Instituto Mexicano del Seguro Social
Other Study IDs: 98337029
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Adrenal Myelolipoma
Keywords: Benign, neoplasms, adrenal myelolipoma
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic adrenalectomy — laparoscopic transabdominal approach.

SUMMARY:
48-year-old woman who presented with intermittent left flank pain with incidental findings of adrenal tumor on computed tomography (CT). She underwent laparoscopic tumor resection due to a large tumor of 12 cm in size.

DETAILED DESCRIPTION:
A 48-year-old female presented to our hospital with the following medical conditions: She denies smoking and drug addiction. Type 2 diabetes mellitus under treatment with metfomin, surgical history of abdominal hysterectomy and open cholecystectomy.

The patient started experiencing pain located in the left flank for 2 months, which was intermittent, yielded to the administration of analgesics, she denied hematuria and weight loss.

On physical examination, the abdomen was distended due to adipose tissue, normal bowel sounds were auscultated, and abdominal masses are not palpable.

She underwent a computed tomography (CT) scan. CT features in the anatomical site of the left adrenal gland, a well-defined ovoid tumor is observed, with heterogeneous content with areas of hypodense (5 HU), fat and calcification. It measures 90 x 69 x 92 mm. Upon application of contrast medium, the hypodense parts present enhancement up to 44 HU. (Fig. 1, 2). She was decided for surgical resection of the tumor via laparoscopic transabdominal approach. The surgery went well without any intraoperative and postoperative complications. She was discharged after day 3.

ELIGIBILITY:
Inclusion Criteria:

* Patient with myelolipoma

Exclusion Criteria:

* Patient without myelolipoma

Min Age: 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 48 Year old Female
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Cure of the disease | 3 days
  Complete myelolipoma resection

CONTACTS AND LOCATIONS:
Locations (1):
- Mexican Institute Of Social Health, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: Yes
manuscript publication
Supporting Information: CSR
Time Frame: July 2024 for ever